CLINICAL TRIAL: NCT03665662
Title: Effect of Intra-procedure Music on Anxiety for Interventional Radiology Procedures
Brief Title: Effect of Intra-procedure Music on Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-01156
Record Dates: First submitted 2018-08-22; First posted 2018-09-11 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in this arm will receive patient-selected music through headphones throughout their procedure.
  Interventions: Other: Music
- Control (No Intervention): Patients will be wearing headphones during their procedure (for the purpose of blinding the care team), but will not receive any music, sounds or sound-cancelling effects through the headphones.

INTERVENTIONS:
Other: Music — Intra-procedure music through headphones
  Arms: Intervention

SUMMARY:
The purpose of this study is to examine the effects of intra-procedure music intervention on procedural anxiety, physiological stress and sedation requirements in patients undergoing moderate sedation procedures. Study participants will be randomly assigned into two groups: 1. Control - standard care without music intervention. 2. Intervention - standard of care plus music intervention. The State-Trait Anxiety Inventory questionnaire will be provided pre, intra and post procedure to all subjects in addition to an exit survey.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old) patients
* Scheduled for moderate sedation procedures in the Interventional Radiology department at Tisch Hospital, NYU Langone Health in New York, New York
* Able to read and write in English at a sixth grade level (STAI is written at sixth grade comprehension level)

Exclusion Criteria:

* Not a moderate sedation candidate (hemodynamically unfit, not optimized for procedure, pregnant)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) score | Up to 12 months
  To examine the effects of intra-procedure music on subjects' anxiety surrounding (pre, during, post) procedures in interventional radiology. Anxiety will be measured by a validated questionnaire called the State-Trait Anxiety Inventory (STAI)

SECONDARY OUTCOMES:
Heart rate | Up to 12 months
  To examine the effects of intra-procedure music on subjects' heart rate in interventional radiology procedures
Respiration rate | Up to 12 months
  To examine the effects of intra-procedure music on subjects' respiration rate in interventional radiology procedures
Blood pressure | Up to 12 months
  To examine the effects of intra-procedure music on subjects' blood pressure in interventional radiology procedures
Amount of sedation required | Up to 12 months
  To examine the effects of intra-procedure music on the amount of sedation required for subjects in interventional radiology procedures
Pain score | Up to 12 months
  To examine the effects of intra-procedure music on the subjects' pain scores during interventional radiology procedures
RASS score | Up to 12 months
  To examine the effects of intra-proceudre music on the subjects' RASS scores during interventional radiology procedures

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horwitz, MD, MHS, Principal Investigator — NYU Langone Health
Locations (1):
- Institutional Review Board Operations (IRB), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No